CLINICAL TRIAL: NCT02382978
Title: Feasibility Study of Nurse-Provided Well Child Care in Family Health Team in Ontario, Canada
Brief Title: Feasibility Study of Nurse-Provided Well Child Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Bruyère Health Research Institute. (Other); College of Family Physicians of Canada (Other); University of Ottawa (Other)
Responsible Party: Principal Investigator, Jolanda Turley, Staff Physician, Associate Professor, MD CCFP, Ottawa Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20150037-01H
Record Dates: First submitted 2015-02-20; First posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Well Child Care; Multidisciplinary Care; Family Medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nurse-provided well child care visit (Experimental): these children will be seen by a nurse only for their regular, pre-scheduled well child care visit
  Interventions: Other: nurse-provided well child visit

INTERVENTIONS:
Other: nurse-provided well child visit

SUMMARY:
This study will test whether or not nurses can provide well child care in a multi-disciplinary primary health care team without physicians also seeing the children at pre-scheduled well child care visits.

DETAILED DESCRIPTION:
This study will deploy a mixed-methods convergent parallel design19, using quantitative methods as well as qualitative data gathering and analyses. To test the acceptability and satisfaction of the care received, interviews with patients and health care team members will investigate attitudes and experiences of patients and care providers. To explore the effectiveness and efficiency of nurse-led WCC, interviews and chart audits will assess the quality of care provided, and costs in terms of time and team resources involved. These two methods will occur simultaneously and the results will be integrated and reported together to give an overall view of the feasibility of nurse-provided WCC within the Bruyere/Primrose FHT.

Sample: There will be 2 cohorts of participants. The first cohort will consist of the health care professionals involved, namely the family physicians and nurses from the Bruyere/Primrose FHT who agree to participate and whose patients will be invited to join the research study. The second cohort of participants will consist of parents of well children who will be asked to have a nurse provide WCC during the pilot project. The eligibility criteria will include:

* Most responsible provider agrees to appropriateness for inclusion
* born at term and from uncomplicated pregnancy and birth
* normal physical growth and development to date
* no parental post-partum depression
* aged between 6 weeks and 4 years of age
* due for WCC visits in the study period Recruitment: The appointment schedules and panels of participating FHT physicians will be reviewed to identify eligible children due or scheduled for a visit. The potential participants will be contacted by phone 1-4 weeks prior to their visit, by the research assistant, and have the project explained to them with an invitation to participate or continue with their usual care. If a parent agrees, verbal informed consent over the phone will be obtained. Consenting patients will be offered the nurse intervention on arrival for their scheduled appointment, with the option of seeing their family physician afterwards. They will sign an informed consent form prior to the visit, which will also ask for interest in participating in follow-up interviews.

Intervention: A proposed work-flow model for nurse-led WCC will be developed, informed by both the literature review and competency-mapping exercise as well as with discussions with the participating FHT physicians and nurses to ensure feasibility and buy-in. It is very likely that the nurses will use the Rourke Baby Record, a standardized and validated template for well child visits, endorsed for use by the College of Family Physicians of Canada20, and used by many physicians at the Bruyere/Primrose clinics. FHT team members of all disciplines will be asked to review the work-flow model during a consultation session to provide feedback, buy-in, and validation. The plan will then be tested with a selected cohort of infants and children and adjustments will be made according to feedback and previously unanticipated issues. The pilot project will then commence and run for a 9-month period to allow for multiple visits with the same patients, recall of patients requiring specific WCC tasks and possibly alternating visits with the nurse and the family physician. The goal is to perform 50 nurse WCC visits within the study period.

Data collection: To address our secondary research question, semi-structured interviews will explore the acceptability of nurse-provided WCC for parents, nurses and physicians at the Bruyere/Primrose FHT, focusing on potential facilitators and barriers to the introduction of such a model of care. Interviews will be held with the provider cohort before and after the intervention phase, and with patients after the nurse WCC visit. Interviews will stopped when theme saturation is achieved or 10 providers and 20 patients have been interviewed, which ever comes first. The interview guide will be developed by the research team using information from the literature review, the competency mapping-exercise and the consultations with the FHT members around recruitment and work-flow planning (see Appendix B for potential interview questions). To further assess the acceptability and feasibility of nurse led WCC, the investigators will compile initial participation rates (percentage of patients contacted who accepted the nurse WCC) and continuation rates (percentage of participants who were eligible for additional visits and who agree to at another nurse-led WCC visit within the study period).

In order to provide quantitative data about the acceptability of nurse-provided WCC, the electronic medical records of participants at the Bruyere/Primrose FHT will be searched for quality indicators such as immunization rates, WCC visits attended by eligible patients, the use of standard developmental questionnaires (eg. the Nippissing District Developmental Screen), the completion of a template like the Rourke Baby Record, the proper documentation of growth parameters, the frequency of visits during the study period, and appropriate follow-up plans according to the WCC visit findings. Further or different indicators may be selected, based on the competency-mapping exercise currently underway. Using the same data extraction sheet developed for the participants' chart audit, similar data will be extracted from a randomly selected age-matched cohort of control subjects not offered the intervention and compared for the nine months before the intervention and during the 9 month study period.

Analyses: The transcripts of the semi-structured interviews will be anonymized and then read by several members of the research team, including the investigators. A coding template will be developed based on the literature review and study objectives and may be iteratively adapted during the initial interviews to allow for emerging themes. Thematic analysis will be used to code the data, at first creating many codes, which will then be grouped and collapsed into major themes and sub-themes21. At analysis meetings, the entire research team will review the codes, themes and sub-themes to reach consensus about how the data answers the question of feasibility and acceptability of nurse-provided WCC. To ensure rigour, these themes will be compared to findings from the literature review and chart audit, triangulated and then, final conclusions will be drawn22, 23, 24.

Quantitative data from the chart audit will be analyzed using SPSS 21 and descriptive statistics will be generated to compare proportions receiving recommended care across the two groups pre- and post-intervention. Our hypothesis is that there will be no difference in the appropriate care manoeuvres received between the control group and the intervention group. Patient characteristics will be summarized and reported by group. Discrete variables will be summarized using frequencies and proportions. Comparisons of discrete variables between groups will be made by using Chi-square or Fisher's exact test, as appropriate. As this is a pilot project, the investigators do not expect to be powered to detect a significant difference in care but these results will be used to triangulate the findings from the qualitative data about appropriate care.

Participation rates will be calculated based on the proportion of invited patients who participate in the intervention. Completion rates will be calculated to determine what proportion of those who start with nurse-provided WCC continue with the intervention for all of their visits during the full duration of the study.

Results: The quantitative and qualitative results will be integrated and reported together to provide a description on the feasibility and acceptability, as well as the efficacy compared to usual care of nurse-provided WCC.

ELIGIBILITY:
Inclusion Criteria:

* Most responsible provider agrees to appropriateness for inclusion
* born at term and from uncomplicated pregnancy and birth
* normal physical growth and development to date
* no parental post-partum depression
* aged between 6 weeks and 4 years of age
* due for WCC visits in the study period

Exclusion Criteria:

-

Ages: 6 Weeks to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-01 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
nurse-provided well child care | 9 months
  qualitative data from interviews and focus groups about acceptability